CLINICAL TRIAL: NCT05266586
Title: A Placebo-Controlled, Double-Blind, Randomized, Phase 2 Study to Evaluate the Effect of Obicetrapib 10 mg Daily in Combination With Ezetimibe 10 mg Daily as an Adjunct to High-Intensity Statin Therapy: The ROSE 2 Study
Brief Title: Study to Evaluate the Effect of Obicetrapib in Combination With Ezetimibe as an Adjunct to HIS Therapy
Acronym: ROSE2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NewAmsterdam Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TA-8995-202
Record Dates: First submitted 2022-02-23; First posted 2022-03-04 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2022-10

CONDITIONS: Dyslipidemias; High Cholesterol; Hypercholesterolemia
Keywords: obicetrapib; statin; LDL-C; cholesterol; atherosclerosis
MeSH Terms: conditions — Dyslipidemias; Hypercholesterolemia; Atherosclerosis | interventions — Ezetimibe

STUDY DESIGN:
Intervention Model Description: Placebo-controlled, double-blind, randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: placebo tablet made to resemble active; placebo capsule made to resemble active
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): once-daily placebo tablet and placebo capsule
  Interventions: Other: Obicetrapib placebo; Other: Ezetimibe placebo
- monotherapy (Experimental): once-daily obicetrapib 10 mg tablet and placebo capsule
  Interventions: Drug: Obicetrapib; Other: Ezetimibe placebo
- combination therapy (Experimental): once-daily obicetrapib 10 mg tablet and ezetimibe 10 mg capsule
  Interventions: Drug: Obicetrapib; Drug: Ezetimibe 10mg

INTERVENTIONS:
Drug: Obicetrapib — tablets
  Other Names: CETP inhibitor
  Arms: combination therapy; monotherapy
Drug: Ezetimibe 10mg — capsules; 10 mg ezetimibe tablets filled into capsule shells, 1 tablet per capsule.
  Arms: combination therapy
Other: Obicetrapib placebo — tablets; no active ingredient
  Arms: Placebo
Other: Ezetimibe placebo — capsules; no active ingredient
  Arms: Placebo; monotherapy

SUMMARY:
This study will be a placebo-controlled, double-blind, randomized, phase 2 study to evaluate the efficacy, safety, and tolerability of obicetrapib 10 mg, both in combination with ezetimibe 10 mg and as monotherapy, as an adjunct to high-intensity statin therapy.

DETAILED DESCRIPTION:
This study will be a placebo-controlled, double-blind, randomized, phase 2 study to evaluate the efficacy, safety, and tolerability of obicetrapib 10 mg, both in combination with ezetimibe 10 mg and as monotherapy, as an adjunct to high-intensity statin therapy. The screening period for this study will take up to 2-weeks. Afterwards patients will be randomized to placebo, 10 mg obicetrapib monotherapy, or 10 mg obicetrapib + 10 mg ezetimibe combination therapy for a 12-week treatment period. After the treatment period, patients will continue for a 4-week safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

* LDL-C > 70 mg/dL and Triglycerides < 400 mg/dL,
* Treated with a high-intensity statin therapy

Exclusion Criteria:

* BMI >= 40 kg/m2
* Significant cardiovascular disease
* HbA1c >= 10%
* Uncontrolled hypertension
* Active muscle disease
* estimated glomerular filtration rate < 60 mL/min
* Hepatic dysfunction
* History of participation in any clinical trial evaluating obicetrapib
* Anemia
* History of malignancy
* Alcohol abuse
* Treatment with investigational product
* Treatment with PCSK9
* Clinically significant condition
* Known CETP inhibitor allergy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2022-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Ditmarsch, Study Director — NewAmsterdam Pharma
Locations (16):
- United States (16):
  - Velocity Clinical Research - Westlake d.b.a National Research Institute, Los Angeles, California
  - Valley Clinical Trials, Inc., Northridge, California
  - Ocala Cardiovascular Research, Ocala, Florida
  - A & R Research Group, LLC, Pembroke Pines, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Meridian Clinical Research - Savannah, GA, Savannah, Georgia
  - Velocity Clinical Research, Meridian, Idaho
  - Biofortis, Inc, Addison, Illinois
  - Northwest Heart Clinical Research, LLC, Arlington Heights, Illinois
  - Midwest Institute for Clinical Research, Indianapolis, Indiana
  - Research Integrity LLC, Owensboro, Kentucky
  - Oakland Medical Research Center, Troy, Michigan
  - Mercury Street Medical, Butte, Montana
  - Meridian Clinical Research- Springdale, OH, Cincinnati, Ohio
  - Aventiv Research, Inc., Columbus, Ohio
  - Summit Research Group, LLC, Munroe Falls, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 231 participants were screened; out of 231, 119 participants were randomized.
Period: Overall Study
Arm/Group | Placebo | Monotherapy | Combination Therapy
Started | 40 | 39 | 40
Completed | 36 | 36 | 38
Not Completed | 4 | 3 | 2
Not completed — Adverse Event | 2 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Non-compliance with study drug | 0 | 1 | 0
Not completed — Subject unable to adhere to all protocol requirements | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Population is defined as all participants who received at least one dose of study drug and had a baseline value for LDL-C assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Monotherapy | Combination Therapy | Total
Number analyzed (Participants) | 40 | 26 | 31 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (8.46) | 64.8 (7.24) | 63.5 (9.08) | 62.6 (8.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 9 | 12 | 35
  Male | 26 | 17 | 19 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 3 | 9
  Not Hispanic or Latino | 35 | 24 | 28 | 87
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 9 | 3 | 2 | 14
  White | 30 | 23 | 29 | 82
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Baseline Low-Density Lipoprotein Cholesterol (LDL-C) Values [Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)] — Baseline LDL-C is defined as the last measurement prior to the first dose of study drug. LDL-C was calculated using the Friedewald Formula.
  milligrams per deciliter (mg/dL) | 99.1 (27.06) | 100.6 (33.65) | 96.0 (25.62) | 98.57 (28.78)

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) for Combination Treatment Group Compared With the Placebo Group [Friedewald]
Description: Mean percent change from Day 1 to Day 84 in Low-Density Lipoprotein Cholesterol (LDL-C) for the obicetrapib 10 mg + ezetimibe 10 mg combination treatment group compared with the placebo group. LDL-C was calculated using the Friedewald equation unless TG
  ≥400 mg/dL or LDL-C ≤50 mg/dL; if TG ≥400 mg/dL or LDL-C ≤50 mg/dL, then LDL-C level was measured directly by preparative ultracentrifugation (PUC).
Time Frame: 12-weeks
Population: On-treatment defined as all randomized participants who received at least 1 dose of any study drug and had a baseline value for low-density lipoprotein cholesterol (LDL-C), excluding those with PK evidence suggesting participant misconduct, i.e., plasma obicetrapib < 100 ng/mL
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Placebo | Combination Therapy
Number analyzed (Participants) | 36 | 31
percent change from baseline | -0.83 (24.514) | -59.07 (14.814)
Statistical Analysis 1: Comparison: Placebo vs Combination Therapy; Test type: Superiority; p < .0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -58.38, 95% CI 2-sided [-68.59 to -48.18], Standard Error of Mean 5.138

2. Primary Outcome: Median Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) for Combination Treatment Group Compared With the Placebo Group [Friedewald]
Description: Median percent change from Day 1 to Day 84 in Low-Density Lipoprotein Cholesterol (LDL-C) for the obicetrapib 10 mg + ezetimibe 10 mg combination treatment group compared with the placebo group. LDL-C was calculated using the Friedewald equation unless TG
  ≥400 mg/dL or LDL-C ≤50 mg/dL; if TG ≥400 mg/dL or LDL-C ≤50 mg/dL, then LDL-C level was measured directly by preparative ultracentrifugation (PUC).
Time Frame: 12-Weeks
Population: as for outcome 1
Measure: Median (Full Range); unit: percent change from baseline
Arm/Group | Placebo | Combination Therapy
Number analyzed (Participants) | 36 | 31
percent change from baseline | -6.35 [-36.4 to 96.7] | -63.40 [-83.7 to -29.7]
Statistical Analysis 1: Comparison: Placebo vs Combination Therapy; Test type: Superiority; p < .0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -58.38, 95% CI 2-sided [-68.59 to -48.18], Standard Error of Mean 5.138

3. Primary Outcome: LS Mean Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) for Combination Treatment Group Compared With the Placebo Group [Friedewald]
Description: LS Mean percent change from Day 1 to Day 84 in Low-Density Lipoprotein Cholesterol (LDL-C) for the obicetrapib 10 mg + ezetimibe 10 mg combination treatment group compared with the placebo group. LDL-C was calculated using the Friedewald equation unless TG
  ≥400 mg/dL or LDL-C ≤50 mg/dL; if TG ≥400 mg/dL or LDL-C ≤50 mg/dL, then LDL-C level was measured directly by preparative ultracentrifugation (PUC).
Time Frame: 12-Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Combination Therapy
Number analyzed (Participants) | 40 | 31
percent change from baseline | -0.85 (3.472) | -59.23 (3.786)
Statistical Analysis 1: Comparison: Placebo vs Combination Therapy; Test type: Superiority; p < .0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -58.38, 95% CI 2-sided [-68.59 to -48.18], Standard Error of Mean 5.138

4. Primary Outcome: Mean Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) for Combination Treatment Group Compared With the Placebo Group [PUC]
Description: Mean percent change from Day 1 to Day 84 in Low-Density Lipoprotein Cholesterol (LDL-C) for the obicetrapib 10 mg + ezetimibe 10 mg combination treatment group compared with the placebo group. LDL-C level was measured by preparative ultracentrifugation (PUC).
Time Frame: 12-Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Placebo | Combination Therapy
Number analyzed (Participants) | 36 | 31
percent change from baseline | -1.49 (23.762) | -59.51 (15.192)
Statistical Analysis 1: Comparison: Placebo vs Combination Therapy; Test type: Superiority; p < .0001, ANCOVA; Least Squares (LS) Means = -58.15, 95% CI 2-sided [-68.47 to -47.83], Standard Error of Mean 5.195

5. Primary Outcome: Median Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) for Combination Treatment Group Compared With the Placebo Group [PUC]
Description: Median percent change from Day 1 to Day 84 in Low-Density Lipoprotein Cholesterol (LDL-C) for the obicetrapib 10 mg + ezetimibe 10 mg combination treatment group compared with the placebo group. LDL-C level was measured by preparative ultracentrifugation (PUC).
Time Frame: 12-Weeks
Population: as for outcome 1
Measure: Median (Full Range); unit: percent change from baseline
Arm/Group | Placebo | Combination Therapy
Number analyzed (Participants) | 36 | 31
percent change from baseline | -3.95 [-34.3 to 91.8] | -62.80 [-82.3 to -31.0]
Statistical Analysis 1: Comparison: Placebo vs Combination Therapy; Test type: Superiority; p < .0001, ANCOVA; Least Squares (LS) Means = -58.15, 95% CI 2-sided [-68.47 to -47.83], Standard Error of Mean 5.195

6. Primary Outcome: LS Mean Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) for Combination Treatment Group Compared With the Placebo Group [PUC]
Description: LS Mean percent change from Day 1 to Day 84 in Low-Density Lipoprotein Cholesterol (LDL-C) for the obicetrapib 10 mg + ezetimibe 10 mg combination treatment group compared with the placebo group. LDL-C level was measured by preparative ultracentrifugation (PUC).
Time Frame: 12-Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Combination Therapy
Number analyzed (Participants) | 36 | 31
percent change from baseline | -1.54 (3.533) | -59.69 (3.811)
Statistical Analysis 1: Comparison: Placebo vs Combination Therapy; Test type: Superiority; p < .0001, ANCOVA; Least Squares (LS) Means = -58.15, 95% CI 2-sided [-68.47 to -47.83], Standard Error of Mean 5.195

7. Secondary Outcome: Mean Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) for Obicetrapib 10 mg Monotherapy Compared With Placebo [Friedewald]
Description: Mean percent change in Low-Density Lipoprotein Cholesterol (LDL-C) from day 1 to day 84 for obicetrapib 10 mg monotherapy treatment group compared with the placebo group. LDL-C was calculated using the Friedewald equation unless TG ≥400 mg/dL or LDL-C ≤50 mg/dL; if TG ≥400 mg/dL or LDL-C ≤50 mg/dL, then LDL-C level was measured directly by preparative ultracentrifugation (PUC).
Time Frame: 12-weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Placebo | Monotherapy
Number analyzed (Participants) | 36 | 26
percent change from baseline | -0.83 (24.514) | -39.35 (22.602)
Statistical Analysis 1: Comparison: Placebo vs Monotherapy; Test type: Superiority; p < .0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -38.35, 95% CI 2-sided [-49.07 to -27.63], Standard Error of Mean 5.397

8. Secondary Outcome: Median Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) for Obicetrapib 10 mg Monotherapy Compared With Placebo [Friedewald]
Description: Median percent change in Low-Density Lipoprotein Cholesterol (LDL-C) from day 1 to day 84 for obicetrapib 10 mg monotherapy treatment group compared with the placebo group. LDL-C was calculated using the Friedewald equation unless TG ≥400 mg/dL or LDL-C ≤50 mg/dL; if TG ≥400 mg/dL or LDL-C ≤50 mg/dL, then LDL-C level was measured directly by preparative ultracentrifugation (PUC).
Time Frame: 12-Weeks
Population: as for outcome 1
Measure: Median (Full Range); unit: percent change from baseline
Arm/Group | Placebo | Monotherapy
Number analyzed (Participants) | 36 | 26
percent change from baseline | -6.35 [-36.4 to 96.7] | -43.50 [-78.4 to 22.6]
Statistical Analysis 1: Comparison: Placebo vs Monotherapy; Test type: Superiority; p < .0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -38.35, 95% CI 2-sided [-49.07 to -27.63], Standard Error of Mean 5.397

9. Secondary Outcome: LS Mean Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) for Obicetrapib 10 mg Monotherapy Compared With Placebo [Friedewald]
Description: LS Mean percent change in Low-Density Lipoprotein Cholesterol (LDL-C) from day 1 to day 84 for obicetrapib 10 mg monotherapy treatment group compared with the placebo group. LDL-C was calculated using the Friedewald equation unless TG
  ≥400 mg/dL or LDL-C ≤50 mg/dL; if TG ≥400 mg/dL or LDL-C ≤50 mg/dL, then LDL-C level was measured directly by preparative ultracentrifugation (PUC).
Time Frame: 12-Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Monotherapy
Number analyzed (Participants) | 40 | 26
percent change from baseline | -0.85 (3.472) | -39.20 (4.133)
Statistical Analysis 1: Comparison: Placebo vs Monotherapy; Test type: Superiority; p < .0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -38.35, 95% CI 2-sided [-49.07 to -27.63], Standard Error of Mean 5.397

10. Secondary Outcome: Mean Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) for Obicetrapib 10 mg Monotherapy Compared With Placebo [PUC]
Description: Mean percent change in Low-Density Lipoprotein Cholesterol (LDL-C) from day 1 to day 84 for obicetrapib 10 mg monotherapy treatment group compared with the placebo group. LDL-C level was measured by preparative ultracentrifugation (PUC).
Time Frame: 12-Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Placebo | Monotherapy
Number analyzed (Participants) | 36 | 26
percent change from baseline | -1.49 (23.762) | -39.04 (23.456)
Statistical Analysis 1: Comparison: Placebo vs Monotherapy; Test type: Superiority; p < .0001, ANCOVA; Least Squares (LS) Means = -37.21, 95% CI 2-sided [-48.07 to -26.35], Standard Error of Mean 5.465

11. Secondary Outcome: Median Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) for Obicetrapib 10 mg Monotherapy Compared With Placebo [PUC]
Description: Median percent change in Low-Density Lipoprotein Cholesterol (LDL-C) from day 1 to day 84 for obicetrapib 10 mg monotherapy treatment group compared with the placebo group. LDL-C level was measured by preparative ultracentrifugation (PUC).
Time Frame: 12-Weeks
Population: as for outcome 1
Measure: Median (Full Range); unit: percent change from baseline
Arm/Group | Placebo | Monotherapy
Number analyzed (Participants) | 36 | 26
percent change from baseline | -3.95 [-34.3 to 91.8] | -43.55 [-78.4 to 20.4]
Statistical Analysis 1: Comparison: Placebo vs Monotherapy; Test type: Superiority; p < .0001, ANCOVA; Least Squares (LS) Means = -37.21, 95% CI 2-sided [-48.07 to -26.35], Standard Error of Mean 5.465

12. Secondary Outcome: LS Mean Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) for Obicetrapib 10 mg Monotherapy Compared With Placebo [PUC]
Description: LS Mean percent change in Low-Density Lipoprotein Cholesterol (LDL-C) from day 1 to day 84 for obicetrapib 10 mg monotherapy treatment group compared with the placebo group. LDL-C level was measured by preparative ultracentrifugation (PUC).
Time Frame: 12-Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Monotherapy
Number analyzed (Participants) | 36 | 26
percent change from baseline | -1.54 (3.533) | -38.75 (4.166)
Statistical Analysis 1: Comparison: Placebo vs Monotherapy; Test type: Superiority; p < .0001, ANCOVA; Least Squares (LS) Means = -37.21, 95% CI 2-sided [-48.07 to -26.35], Standard Error of Mean 5.465

13. Secondary Outcome: Mean Percent Change in Apolipoprotein-B (ApoB) for Obicetrapib in Combination With Ezetimibe Compared to Placebo
Description: Mean percent change from day 1 to day 84 in Apolipoprotein-B (ApoB) for the obicetrapib 10 mg plus ezetimibe 10 mg combination treatment group compared with the placebo group
Time Frame: 12-weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change from baseline
Groups:
- Combination Therapy: once-daily obicetrapib 10 mg tablet and ezetimibe 10 mg capsule Obicetrapib: tablets Ezetimibe 10mg: capsules; 10 mg ezetimibe tablets filled into capsule shells, 1 tablet per capsule.
Arm/Group | Placebo | Combination Therapy
Number analyzed (Participants) | 36 | 31
percent change from baseline | 0.51 (19.784) | -34.66 (11.796)
Statistical Analysis 1: Comparison: Placebo vs Combination Therapy; Test type: Superiority; p < .0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -35.68, 95% CI 2-sided [-43.23 to -28.13], Standard Error of Mean 3.800

14. Secondary Outcome: Median Percent Change in Apolipoprotein-B (ApoB) for Obicetrapib in Combination With Ezetimibe Compared to Placebo
Description: Median percent change from day 1 to day 84 in Apolipoprotein-B (ApoB) for the obicetrapib 10 mg plus ezetimibe 10 mg combination treatment group compared with the placebo group
Time Frame: 12-Weeks
Population: as for outcome 1
Measure: Median (Full Range); unit: percent change from baseline
Arm/Group | Placebo | Combination Therapy
Number analyzed (Participants) | 36 | 31
percent change from baseline | -2.05 [-30.9 to 76.9] | -34.40 [-54.3 to -14.7]
Statistical Analysis 1: Comparison: Placebo vs Combination Therapy; Test type: Superiority; p < .0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -35.68, 95% CI 2-sided [-43.23 to -28.13], Standard Error of Mean 3.800

15. Secondary Outcome: LS Mean Percent Change in Apolipoprotein-B (ApoB) for Obicetrapib in Combination With Ezetimibe Compared to Placebo
Description: LS Mean percent change from day 1 to day 84 in Apolipoprotein-B (ApoB) for the obicetrapib 10 mg plus ezetimibe 10 mg combination treatment group compared with the placebo group
Time Frame: 12-Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Combination Therapy
Number analyzed (Participants) | 40 | 31
percent change from baseline | 0.72 (2.572) | -34.95 (2.796)
Statistical Analysis 1: Comparison: Placebo vs Combination Therapy; Test type: Superiority; p < .0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -35.68, 95% CI 2-sided [-43.23 to -28.13], Standard Error of Mean 3.800

16. Secondary Outcome: Mean Percent Change in Apolipoprotein-B (ApoB) for Obicetrapib 10 mg Monotherapy Compared With Placebo
Description: Mean percent change from day 1 to day 84 in Apolipoprotein-B (ApoB) for the obicetrapib 10 mg monotherapy treatment group compared with the placebo group
Time Frame: 12-weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Placebo | Monotherapy
Number analyzed (Participants) | 36 | 26
percent change from baseline | 0.51 (19.784) | -21.73 (16.057)
Statistical Analysis 1: Comparison: Placebo vs Monotherapy; Test type: Superiority; p < .0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -22.28, 95% CI 2-sided [-30.21 to -14.36], Standard Error of Mean 3.991

17. Secondary Outcome: Median Percent Change in Apolipoprotein-B (ApoB) for Obicetrapib 10 mg Monotherapy Compared With Placebo
Description: Median percent change from day 1 to day 84 in Apolipoprotein-B (ApoB) for the obicetrapib 10 mg monotherapy treatment group compared with the placebo group
Time Frame: 12-Weeks
Population: as for outcome 1
Measure: Median (Full Range); unit: percent change from baseline
Arm/Group | Placebo | Monotherapy
Number analyzed (Participants) | 36 | 26
percent change from baseline | -2.05 [-30.9 to 76.9] | -24.20 [-44.8 to 27.1]
Statistical Analysis 1: Comparison: Placebo vs Monotherapy; Test type: Superiority; p < .0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -22.28, 95% CI 2-sided [-30.21 to -14.36], Standard Error of Mean 3.991

18. Secondary Outcome: LS Mean Percent Change in Apolipoprotein-B (ApoB) for Obicetrapib 10 mg Monotherapy Compared With Placebo
Description: LS Mean percent change from day 1 to day 84 in Apolipoprotein-B (ApoB) for the obicetrapib 10 mg monotherapy treatment group compared with the placebo group
Time Frame: 12-Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Monotherapy
Number analyzed (Participants) | 40 | 26
percent change from baseline | 0.72 (2.572) | -21.56 (3.052)
Statistical Analysis 1: Comparison: Placebo vs Monotherapy; Test type: Superiority; p < .0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -22.28, 95% CI 2-sided [-30.21 to -14.36], Standard Error of Mean 3.991

ADVERSE EVENTS:
Time Frame: From first dose of study drug through Week 16
Description: The Safety Population was defined as all participants who received at least 1 dose of any study drug.
Arm/Group | Placebo | Monotherapy | Combination Therapy
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/39 | 0/40
Serious Adverse Events (participants affected / at risk) | 1/40 | 1/39 | 0/40
Other Adverse Events (participants affected / at risk) | 16/40 | 8/39 | 11/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=40) | Monotherapy (N=39) | Combination Therapy (N=40)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=40) | Monotherapy (N=39) | Combination Therapy (N=40)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 1 (2)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (3) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After the multicenter publication or 12 months after completion of the study, whichever occurs first, Institution may publish the results of its study data. Institution and PI shall provide sponsor with an advance copy of any proposed communications at least 60 days prior and Sponsor shall have 60 days to review. Sponsor may request (a) the deletion of any Confidential Information, (b) reasonable changes, or (c) a delay for an additional period, not to exceed 90 days.

DOCUMENTS (2):
  • Study Protocol (2021-09-16): https://cdn.clinicaltrials.gov/large-docs/86/NCT05266586/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-20): https://cdn.clinicaltrials.gov/large-docs/86/NCT05266586/SAP_001.pdf